CLINICAL TRIAL: NCT01789424
Title: Valuation of Airway Protection (Swalling) in Patient Sedated for Gastroenteric Endoscopic Procedure
Brief Title: Valuation of Swallowing in Patient Sedated for Gastroenteric Endoscopic Procedure
Acronym: SwallSed
Status: Completed | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Agostoni Massimo, Medical Doctor, Ospedale San Raffaele
Other Study IDs: Swallsed; Swallsed2012
Record Dates: First submitted 2013-01-28; First posted 2013-02-12 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Sedation for Gastroenteric Endoscopic Procedure; Deglutition Disorders; Aspiration of Food
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim of this study is to evaluate swallowing functionality in patient sedated for gastroenteric endoscopic procedure.

Swallowing will be study by laryngeal fibroscopy and evaluate using Penetration-Aspiration Scale and Aspiration Risk validated in scientific literature.

Aim of the study is to describe swallowing, as an expression of airway protection, in sedated patient. in particular, our purpose is to determine the incidence of moderate-severe and severe swallowing alteration (level 3 or 4 of Aspiration Risk scale).

DETAILED DESCRIPTION:
All patients will be sedated using propofol target controlled infusion (TCI) with a target of 2-5 mcg/ml During sedation and examination will be monitored: cardiac frequency, peripheral oxygen saturation and non-invasive arterial blood pressure.

During sedation, before starting the gastroenteric endoscopic exam, will be performed a fibroscopic swallowing evaluation made by an expert otolaryngologist.

Fibroscopic evaluation consist of:

* laryngeal fibroscopy to evaluate vocal cord motility
* swallowing trial using 3 blue colored water bolus (3-4ml) and computing a " Penetration-aspiration scale" and an " Aspiration risk scale"

Rosenbek, Robbins et al. A Penetration-Aspiration Scale. Dysphagia 11:93-98, 1996:

1. No penetration in the airway
2. Bolus reaches the airway, it does not reach vocal cords and it is completely eliminated
3. Bolus reaches the airway, it does not reach vocal cords but it is not completely eliminated
4. Bolus reaches the airway, it reaches vocal cords but it is completely eliminated
5. Bolus reaches the airway, it reaches vocal cords and it is not completely eliminated
6. Bolus reaches the airway, it passes trough vocal cords but it is completely eliminated
7. Bolus reaches the airway, it passes trough vocal cords, it is not eliminated but patient strives to expel it
8. Bolus reaches the airway, it passes trough vocal cords, it is not eliminated and patient does not strive to expel it

Daniels e coll.: Clinical Predictors of Dysphagia and Aspiration Risk: Outcome Measures in Acute Stroke Patients. Arch Phys Med Rehab Vol 81, August 2000:

1. Normal swallowing : no aspiration or penetration in the airway
2. Trivial swallowing impairment: oral or pharyngeal impairment that causes occasional airway penetration with rapid clearance
3. Moderate swallowing impairment: oral or pharyngeal impairment that causes consistent airway penetration with stasis into the vestibule or two or less event of aspiration of a similar viscosity aliment
4. Moderate-severe swallowing impairment: oral or pharyngeal impairment that causes an important aspiration of a similar viscosity aliment
5. Severe swallowing impairment: oral or pharyngeal impairment that causes an important aspiration of similar or different viscosity

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II-III
* Able to give written consent with none exclusion criteria.

Exclusion Criteria:

* presence of feeding tube
* presence of tracheostomy actual or in the past
* severe respiratory deficit
* neurological disease which can compromise swallowing function
* history of surgery for mouth or pharyngeal or esophageal cancer
* history of otolaryngology surgery
* faring-laryngeal radiotherapy
* emergent procedure
* psychic alteration
* patient in therapy with any kind of antidepressant drugs
* insulin dependent diabetes mellitus patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient sedated for gastroenteric endoscopic examination
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Swallowing impairment | 12 months
  Primary outcomes of this study is to verify if there is any kind of swallowing impairment during sedation with propofol and to quantify the eventual impairment.
  Swallowing function will be study by fibroscopic evaluation, that consists of:
  * laryngeal fibroscopy to evaluate vocal cord motility
  * swallowing trial using 3 blue colored water bolus (3-4ml) and computing a " Penetration-aspiration scale" and an " Aspiration risk scale" (see above)

SECONDARY OUTCOMES:
Inhalation | 12 months
  Secondary outcome of this study is to determine if the eventual swallowing impairment during propofol sedation causes inhalation in the airway.
  We use fibroscopic evaluation to identify and to quantify the possible inhalation.
  The fibroscopic evaluation consists of:
  * laryngeal fibroscopy to evaluate vocal cord motility
  * swallowing trial using 3 blue colored water bolus (3-4ml) and computing a " Penetration-aspiration scale" and an " Aspiration risk scale" (see above)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Italy, Italy

REFERENCES:
- [Derived] Gemma M, Pasin L, Oriani A, Agostoni M, Palonta F, Ramella B, Bussi M, Beretta L. Swallowing Impairment During Propofol Target-Controlled Infusion. Anesth Analg. 2016 Jan;122(1):48-54. doi: 10.1213/ANE.0000000000000796. PMID 26049781